CLINICAL TRIAL: NCT06642454
Title: A Randomized Double-Blind Active-Controlled Crossover Trial of Respiratory-Gated Versus Non-Gated Transcutaneous Auricular Vagus Nerve Stimulation for the Treatment of Motor and Non-Motor Symptoms in Parkinson's Disease
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Anhui Medical University (Other)
Responsible Party: Principal Investigator, WANG KAI, Head, Dept of Neurology & Medical Psychology, Director, Cognitive Neuropsychology Lab, PRC, Anhui Medical University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: PD-TaVNS-OPEN
Record Dates: First submitted 2024-10-13; First posted 2024-10-15 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-06

CONDITIONS: Parkinson Disease; Apathy; Sleep Disorder; Motor Disorders; Mood Disorders
MeSH Terms: conditions — Parkinson Disease; Lethargy; Sleep Wake Disorders; Motor Disorders; Mood Disorders

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- 25 Hz non-expiratory gated taVNS (Experimental): 25 Hz non-expiratory gated transcutaneous auricular vagus nerve stimulation
  Interventions: Other: Transcutaneous auricular vagus nerve stimulation
- 25 Hz expiratory gated taVNS (Experimental): 25 Hz expiratory gated transcutaneous auricular vagus nerve stimulation
  Interventions: Other: Transcutaneous auricular vagus nerve stimulation
- 100 Hz expiratory gated taVNS (Experimental): 100 Hz expiratory gated transcutaneous auricular vagus nerve stimulation
  Interventions: Other: Transcutaneous auricular vagus nerve stimulation

INTERVENTIONS:
Other: Transcutaneous auricular vagus nerve stimulation — Stimulation Target: Left cymba conchae.
  25 Hz Non-Expiratory Gated taVNS: Stimulation is delivered for 30 seconds at a frequency of 25 Hz, followed by a 30-second interval.
  25 Hz Expiratory Gated taVNS: One second of stimulation occurs during exhalation at a frequency of 25 Hz.
  100 Hz Expiratory Gated taVNS: One second of stimulation is administered during exhalation at a frequency of 100 Hz.

SUMMARY:
The goal of this clinical trial is to compare the effects of different modes and frequencies of transcutaneous auricular vagus nerve stimulation (taVNS) on motor and non-motor symptoms in people with Parkinson's disease. The main questions it aims to answer are:

Which mode and frequency of taVNS is most effective in improving motor or non-motor symptoms? Are there any side effects or safety concerns with different taVNS frequencies? Researchers will compare three types of taVNS: 25 Hz non-expiratory gated, 25 Hz expiratory gated, and 100 Hz expiratory gated stimulation.

Participants will:

Receive each type of taVNS in three 2-week cycles, with 2-month breaks between cycles Undergo neuropsychological assessments, imaging, eye-tracking, and biological sample collection before and after each cycle.

DETAILED DESCRIPTION:
This study employs a three-cycle crossover design to compare the effects of three different modes and frequencies of transcutaneous auricular vagus nerve stimulation (taVNS). The interventions include: 25 Hz non-expiratory gated taVNS, 25 Hz expiratory gated taVNS, and 100 Hz expiratory gated taVNS. Participants will be randomly assigned to one of three groups, with each group receiving a different intervention during each cycle, lasting 2 weeks per cycle. A 2-month washout period will be implemented between cycles to eliminate any carryover effects.The study design will include neuropsychological assessments, imaging, eye-tracking data collection, and biological specimen collection before and after each intervention.

ELIGIBILITY:
Inclusion Criteria:

* Age: 40 years or older.
* Confirmed diagnosis of Parkinson's disease (PD) per the United Kingdom Brain Bank Criteria by a neurologist specialized in movement disorders.
* Participants must be on a stable dose of all medications for at least 2 weeks, with no planned adjustments to anti-PD medications for the next 3 months.
* In the second version of the Non-Motor Symptoms Scale (NMSS-2) for Parkinson's disease, a score of ≥1 is assigned to either question 4 or question 8.
* Participants must be in good mental health and capable of completing behavioral tests and transcutaneous auricular vagus nerve stimulation.

Exclusion Criteria:

* Mini-Mental State Examination (MMSE) score <24.
* History of head injury, stroke, or other neurological disorders.
* Includes implanted cardiac pacemakers post-DBS operation, local infections, ear loss, or metal implants at the stimulation site.
* Current use of nonsteroidal anti-inflammatory drugs (NSAIDs) or corticosteroids.
* Inability to complete follow-up assessments.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-10-01 (Actual); Primary Completion 2026-12-01 (Estimated); Study Completion 2027-04-01 (Estimated)

PRIMARY OUTCOMES:
Unified Parkinson's Disease Rating Scale Part III (UPDRS-III) | Baseline;2 weeks; 10 weeks; 12 weeks;20 weeks;22weeks
  The Unified Parkinson's Disease Rating Scale, Part III (UPDRS-III) is the gold standard, clinician-administered motor examination for Parkinson's disease. It is a semi-quantitative scale comprising 18 items assessing core motor features-tremor, rigidity, bradykinesia, and postural/gait dysfunction. Each item is scored from 0 (normal) to 4 (severe), with a total possible score of 108. As the primary endpoint in clinical trials, it objectively quantifies motor disability severity and treatment response.
Non-Motor Symptoms Scale, Second Version (NMSS-2) | Baseline;2 weeks; 10 weeks; 12 weeks;20 weeks;22weeks
  The NMSS-2 is a comprehensive, clinician-administered tool designed to assess the range and severity of non-motor symptoms in individuals with Parkinson's disease. It covers multiple domains including sleep disturbances, mood, cognition, gastrointestinal symptoms, urinary dysfunction, and other non-motor manifestations. This second version of the scale provides an updated and refined assessment framework to capture the broad impact of non-motor symptoms on patients' quality of life.

SECONDARY OUTCOMES:
Apathy Motivation Index (AMI) | Baseline;2 weeks; 10 weeks; 12 weeks;20 weeks;22weeks
  Apathy Motivation Index (AMI) The AMI is used to assess levels of apathy across behavioral, emotional, and cognitive domains. It provides a comprehensive measure of motivation deficits.
Apathy Evaluation Scale (AES) | Baseline;2 weeks; 10 weeks; 12 weeks;20 weeks;22weeks
  The AES is designed to evaluate the severity of apathy in individuals, focusing on the lack of motivation in behaviors, emotional responsiveness, and cognitive functioning.
Fatigue Scale-14 (FS-14) | Baseline;2 weeks; 10 weeks; 12 weeks;20 weeks;22weeks
  The FS-14 is a self-report measure used to evaluate fatigue across physical and mental dimensions. It comprises 14 items that assess the severity and impact of fatigue on daily functioning.
Pittsburgh Sleep Quality Index (PSQI) | Baseline;2 weeks; 10 weeks; 12 weeks;20 weeks;22weeks
  The PSQI is a standardized tool used to assess sleep quality and disturbances over a one-month time interval. It evaluates seven components of sleep, including subjective sleep quality, latency, duration, and daytime dysfunction.
REM Sleep Behavior Disorder Screening Questionnaire (RBDSQ) | Baseline;2 weeks; 10 weeks; 12 weeks;20 weeks;22weeks
  The RBDSQ is a diagnostic tool used to screen for REM Sleep Behavior Disorder (RBD), focusing on the presence of dream-enactment behaviors and other sleep-related symptoms.
Hamilton Anxiety Rating Scale (HAMA) | Baseline;2 weeks; 10 weeks; 12 weeks;20 weeks;22weeks
  The HAMA is a clinician-administered scale designed to assess the severity of anxiety symptoms. It covers both psychological and somatic symptoms, providing a comprehensive evaluation of anxiety levels.
Hamilton Depression Rating Scale (HAMD-17) | Baseline;2 weeks; 10 weeks; 12 weeks;20 weeks;22weeks
  The HAMD-17 is a widely used instrument for assessing the severity of depressive symptoms. It consists of 17 items that evaluate mood, physical symptoms, and cognitive disturbances associated with depression.
Epworth Sleepiness Scale (ESS) | Baseline;2 weeks; 10 weeks; 12 weeks;20 weeks;22weeks
  The Epworth Sleepiness Scale (ESS) is a standardized self-report questionnaire measuring daytime sleep propensity. It lists eight common situations; respondents rate their likelihood of dozing (0-3) in each. The total score (0-24) quantifies subjective daytime sleepiness. It is a widely used screening tool for sleep disorders and treatment assessment.

CONTACTS AND LOCATIONS:
Locations (1):
- Cognitive Neuropsychology Lab Anhui Medical University, Hefei, Anhui, China

IPD SHARING:
Plan to Share IPD: No